CLINICAL TRIAL: NCT06596512
Title: Improving the Quality of Care for Asthma Patients at Risk of Exacerbations
Acronym: iCARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Elliot Israel, MD, Professor of Medicine Harvard Medical School Gloria M. and Anthony C. Simboli Distinguished Chair in Asthma Research Director of Clinical Research Pulmonary and Critical Care Division Allergy and Immunology Brigham & Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024P001955
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Moderate-to-Severe Asthma
Keywords: ICS reliever therapy, Decrease exacerbations, iCARE

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PARTICS - Non Frequent Nebulizer Users (Active Comparator): Participants who use a nebulizer less than once a week are Non Frequent Nebulizer (NFN) Users. Adding the PARTICS strategy - Patient Activated Reliever-Triggered Inhaled CorticoSteroid (PARTICS). Patient will use inhaled corticosteroid at time of reliever inhaler or after reliever nebulizer use.
  Interventions: Drug: PARTICS using a single ICS add on
- PARTICS - Frequent Nebulizer User (Active Comparator): Participants who use a nebulizer once a week or more are "Frequent Nebulizer Users". Addition of the PARTICS strategy - Patient Activated Reliever-Triggered Inhaled CorticoSteroid (PARTICS). Patient will use inhaled corticosteroid at time of rescue inhaler or rescue nebulizer use
  Interventions: Drug: PARTICS using a single ICS add on
- MART (non frequent nebulizer users) - MART strategy - Maintenance and Reliever Therapy (Active Comparator): Participants who use a nebulizer less than once a week are Non Frequent Nebulizer (NFN) Users. MART strategy is a ICS/LABA combination therapy for maintenance and relief.
  Interventions: Drug: MART
- MART (frequent nebulizer users) (Active Comparator): Participants who use a nebulizer once a week or more are Frequent Nebulizer Users. MART strategy is a ICS/LABA combination therapy for maintenance and relief.
  Interventions: Drug: MART

INTERVENTIONS:
Drug: PARTICS using a single ICS add on — Participants randomized to PARTICS who use a nebulizer less than once a week are instructed to use the study prescribed ICS each time they use their rescue inhaler and take 5 puffs of the newly prescribed ICS after each rescue nebulizer use.
  Other Names: Patient Activated Reliever Triggered ICS
  Arms: PARTICS - Frequent Nebulizer User; PARTICS - Non Frequent Nebulizer Users
Drug: MART — Participants are instructed to use prescribed study ICS/LABA for maintenance and as needed for rescue.
  Arms: MART (frequent nebulizer users); MART (non frequent nebulizer users) - MART strategy - Maintenance and Reliever Therapy

SUMMARY:
The goal of this trial test two known effective asthma strategies. Treatment guidelines recommend combination therapy of inhaled corticosteroids (ICS) with a long-acting beta-agonist (LABA) inhaled medications. This strategy is known as MART (maintenance and reliever therapy). The second strategy is PARTICS (patient activated reliever triggered ICS) strategy instructs patients to use an ICS metered dose inhaler (ICS) each time they use their rescue inhaler. In addition, they are instructed to take 5 puffs of the ICS after each rescue nebulizer use. PARTICS has been shown to reduce exacerbations, increase asthma control and quality of life, however, the question remains if PARTICS is as effective as MART and therefore be an alternative to MART. This trial will test PARTICS and MART head-to-head.

The trial will include adults with moderate-to-severe asthma at risk for an asthma exacerbation, currently using a combination ICS.

The main questions aim to answer:

* Is PARTICS as effective as SMART?
* Might PARTICS be more effective than SMART? Is the relative effectiveness of PARTICS versus SMART affected by frequent nebulizer use for asthma relief?
* Do PARTICS and SMART diverge in terms of their effectiveness on differing asthma outcomes important to patients?
* Do socioeconomic factors affect the relative effectiveness of PARTICS and SMART? Researchers will compare non frequent nebulizer (NFN) users - less than once a week to frequent nebulizer users - once a week or more, to assess whether the PARTICS strategy is ono-inferior (or superior to the MART strategy in reducing exacerbations, (primary outcome), increasing asthma control and quality of life and decrease days lost from work/school or usual activities.

Most participants will be consented, enrolled, and randomized virtually, others will be consented, enrolled and randomized in person. Once randomized they will be instructed on how to use the prescribed medication:

* Participants randomized to MART will be instructed to use the prescribed ICS/LABA for maintenance and as needed for rescue.
* Participants randomized to PARTICS will be instructed to use the prescribed ICS each time they use their rescue inhaler and take 5 puffs of the newly prescribed ICS after each rescue nebulizer use.
* Participants will be followed for 16 months by monthly survey.

DETAILED DESCRIPTION:
Asthma affects 25 million people in the USA with a disproportionate effect on African American/Black (AA/B) and Hispanic/Latinx (H/L) patients. Inhaled corticosteroids are the backbone of asthma therapy. A so-called SMART (Single Maintenance And Reliever Therapy) approach to ICS therapy has been recommended by US and international guidelines for patients with moderate to severe asthma, because it has been shown in multiple studies to reduce asthma exacerbations. However, these studies have been explanatory, with narrow entry criteria, have only been performed ex- US (with a formulation not available in the US), and have not included significant numbers of AA/B and H/L patients.

Further, there are significant barriers to implementation which include those related to patient patterns of concomitant medication use and beliefs. In a PCORI-funded pragmatic study in 1200 AA/B and H/L patients with asthma, designed with patient partners, we studied an alternative approach we call PARTICS (Patient Activated Reliever Triggered ICS). We reported, in this study published in the New England Journal of Medicine in 2022, that we not only reduced asthma exacerbations, we also improved other outcomes important to patients including asthma control, quality of life and days lost from school, work or usual activities. Our patient advisors have published on their positive experience and other advisors have collaborated with us to publish 9 additional papers which include such topics as an exploration of how socioeconomic factors affect asthma outcomes and how to simply identify patients at risk for asthma exacerbations, among additional topics. Both SMART and PARTICS have advantages and drawbacks. As seen in letters of support from the heads of the US and international guidelines for asthma treatment committees, the lack of direct comparison between the two represents a major gap in knowledge required to formulate best-care practice recommendations.

Specifically, it is unclear as to what degree one approach can substitute for the other and whether they differentially affect distinct domains of asthma outcomes. In collaboration with our advisors, we therefore propose iCARE (Improving the Quality of Care for Asthma patients at Risk of Exacerbations), a large pragmatic study to directly compare SMART to PARTICS in diverse populations and across multiple domains. The study results, regardless of outcome, will help guide the approach to patient-centered asthma care.

ELIGIBILITY:
Inclusion Criteria:

* Clinician diagnosis of asthma for ≥1 year;
* Age at enrollment--18-75 years old inclusive;
* One or more AEXs that occurred < 12 months prior to enrollment. An AEX is defined as an asthma deterioration that either requires 72 hours or more of an oral or parenteral steroids OR a hospital stay for more than 24 hours for asthma. In the case of patients on biologics for asthma, the exacerbation must have also occurred after at least 6 months of biologic therapy;
* Currently prescribed an ICS/LABA containing preparation containing at least the lowest dose of ICS described in Table 2 as regular daily maintenance therapy for at least one month;
* Has a rescue SABA containing inhaler that they have used on average at least once a month.
* Able to provide consent in English for the feasibility study or in English or Spanish for the full study.

Exclusion Criteria:

* Life expectancy <2 years;
* COPD diagnosis unless: a) they were a never smoker; OR b) former smoker with normal pulmonary function tests (PFT; FEV1/FVC ratio of >70%); OR c) current smoker with normal PFTs within 24 months of enrollment; OR d) current or former smoker with obstruction on PFTs (FEV1/FVC ratio of <70% but who demonstrates BOTH >12% acute bronchodilator reversibility AND a normal diffusing capacity both within 24 months of enrollment (criteria successfully used in PREPARE);
* Use of single inhaler product that contains an ICS, LAMA and LABA or one containing both LABA and LAMA within 1 month of enrollment;
* Use of current biologic for less than 6 months;
* Known allergy to any of the components of the intervention;
* Coexisting lung disease (e.g. Cystic Fibrosis, connective tissue disease (unless asthma preceded diagnosis of connective tissue disease by at least 2 years), prematurity-born at 32 weeks or sooner, organ transplantation, bronchiectasis, sarcoid, and obliterative bronchiolitis, among others)
* Has been in an asthma drug treatment trial in past 60 days or within 5 half-lives, whichever is longer, prior to study visit.
* Living in household with someone already enrolled in the study.
* Using daily or every other day oral corticosteroids for asthma or any other condition
* An AEX in the prior 4 weeks
* History of bronchial thermoplasty in prior 6 months
* Poorly or uncontrolled atrial fibrillation
* Not on stable asthma medications for at least 1 month prior to enrollment
* Using doses of ICS/LABA lower than the minimum below:
* Budesonide 320 ug,
* Fluticasone Advair Diskus/ Wixela 200-250 ug Advair HFA 180-230ug Airduo 110-113 ug Breo 100 ug
* Mometasone 200 ug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4100 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Exacerbations | Exacerbation information will be collected via monthly survey for 16 months.
  The primary outcome is annualized rate of asthma exacerbations, defined as 72 hours of parenteral or oral corticosteroids to treat asthma symptoms or an asthma related-hospitalization. Participants are asked on their monthly surveys if they have had an exacerbation requiring at least 3 days of oral steroids or a hospitalization. If the participant answers yes to these questions, the clinical coordinating center contacts the site study coordinator to confirm an exacerbation in the patients EHR. If there is no record of an exacerbation in the EHR, the CCC contacts the patient for details. The information is entered into an exacerbation database and is reviewed separately by two investigators. If they are in agreement, the outcome is recorded (exacerbation yes or exacerbation no). If they do not agree or are unable to definitively determine if the patient had an exacerbation or not, the information goes to the adjudication committee of 3 for determination.

SECONDARY OUTCOMES:
Asthma Control over time | Monthly for 16 months
  Asthma control represents the degree to which impairment (impact of asthma on patient's daily life) is minimized and the goals of therapy are met. The Asthma Control Test is a participant-administered tool for assessing the level of asthma control. Total scores range from 5 to 25, with a score of 20 to 25 indicating well-controlled asthma, a score of 16 to 19 indicating asthma that was not well controlled, and a score of 5 to 15 indicating very poorly controlled asthma. The minimal clinically important difference is 3 points
Asthma Symptom Utility Index (ASUI), Preference based quality of life | Monthly for 16 months
  The ideal outcome measure for any comparative effectiveness analysis captures the risks and benefits for each of the interventions from the patient's point of view. The use of a preference-based instrument, the Asthma Symptom Utility Index (ASUI), captures this important information. The Asthma Symptom Utility Index is a participant-administered tool for assessing preference-based quality of life. Scores range from 0 (worst possible symptoms) to 1 (no symptoms). The minimal clinically important difference is 0.09.
Days Lost Per Year From School/Work or Usual Activities | Monthly for 16 months
  Defined as days not able to work or go to school because of asthma symptoms OR days not able to carry out usual activities due to asthma

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Yale University, New Haven, Connecticut
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data and data dictionary.
Time Frame: The IPD will be available one year after the final research report is posted by our funder, PCORI which has not yet been determined.
Access Criteria: As required by the funder, the data and supporting information will be submitted to the University of Michigan, hosts of the Inter-University Consortium for Pollical and Social Research. Researchers will submit a request to ICPSR and go through a vetting process for approval to receive the data and supporting documents.
URL: https://www.icpsr.umich.edu/web/pages/

REFERENCES:
- [Background] Israel E, Cardet JC, Carroll JK, Fuhlbrigge AL, Pace WD, Maher NE, She L, Rockhold FW, Fagan M, Forth VE, Hernandez PA, Manning BK, Rodriguez-Louis J, Shields JB, Coyne-Beasley T, Kaplan BM, Rand CS, Morales-Cosme W, Wechsler ME, Wisnivesky JP, White M, Yawn BP, McKee MD, Busse PJ, Kaelber DC, Nazario S, Hernandez ML, Apter AJ, Chang KL, Pinto-Plata V, Stranges PM, Hurley LP, Trevor J, Casale TB, Chupp G, Riley IL, Shenoy K, Pasarica M, Calderon-Candelario RA, Tapp H, Baydur A. A randomized, open-label, pragmatic study to assess reliever-triggered inhaled corticosteroid in African American/Black and Hispanic/Latinx adults with asthma: Design and methods of the PREPARE trial. Contemp Clin Trials. 2021 Feb;101:106246. doi: 10.1016/j.cct.2020.106246. Epub 2020 Dec 11. PMID 33316456
- [Background] Expert Panel Working Group of the National Heart, Lung, and Blood Institute (NHLBI) administered and coordinated National Asthma Education and Prevention Program Coordinating Committee (NAEPPCC); Cloutier MM, Baptist AP, Blake KV, Brooks EG, Bryant-Stephens T, DiMango E, Dixon AE, Elward KS, Hartert T, Krishnan JA, Lemanske RF Jr, Ouellette DR, Pace WD, Schatz M, Skolnik NS, Stout JW, Teach SJ, Umscheid CA, Walsh CG. 2020 Focused Updates to the Asthma Management Guidelines: A Report from the National Asthma Education and Prevention Program Coordinating Committee Expert Panel Working Group. J Allergy Clin Immunol. 2020 Dec;146(6):1217-1270. doi: 10.1016/j.jaci.2020.10.003. PMID 33280709
- [Background] Reddel HK, Bacharier LB, Bateman ED, Brightling CE, Brusselle GG, Buhl R, Cruz AA, Duijts L, Drazen JM, FitzGerald JM, Fleming LJ, Inoue H, Ko FW, Krishnan JA, Levy ML, Lin J, Mortimer K, Pitrez PM, Sheikh A, Yorgancioglu AA, Boulet LP. Global Initiative for Asthma Strategy 2021: Executive Summary and Rationale for Key Changes. J Allergy Clin Immunol Pract. 2022 Jan;10(1S):S1-S18. doi: 10.1016/j.jaip.2021.10.001. Epub 2021 Oct 28. PMID 34718211
- [Background] Imam SF, Zafar S, Oppenheimer JJ. Single maintenance and reliever therapy in treatment of asthma exacerbations. Ann Allergy Asthma Immunol. 2022 Dec;129(6):703-708. doi: 10.1016/j.anai.2022.07.024. Epub 2022 Jul 29. PMID 35914659
- [Background] Sobieraj DM, Weeda ER, Nguyen E, Coleman CI, White CM, Lazarus SC, Blake KV, Lang JE, Baker WL. Association of Inhaled Corticosteroids and Long-Acting beta-Agonists as Controller and Quick Relief Therapy With Exacerbations and Symptom Control in Persistent Asthma: A Systematic Review and Meta-analysis. JAMA. 2018 Apr 10;319(14):1485-1496. doi: 10.1001/jama.2018.2769. PMID 29554195
- [Background] Patel M, Pilcher J, Pritchard A, Perrin K, Travers J, Shaw D, Holt S, Harwood M, Black P, Weatherall M, Beasley R; SMART Study Group. Efficacy and safety of maintenance and reliever combination budesonide-formoterol inhaler in patients with asthma at risk of severe exacerbations: a randomised controlled trial. Lancet Respir Med. 2013 Mar;1(1):32-42. doi: 10.1016/S2213-2600(13)70007-9. Epub 2013 Mar 4. PMID 24321802